CLINICAL TRIAL: NCT05361330
Title: A Multicenter Clinical Study to Evaluate the Efficacy and Safety of Shuganjieyu Capsule Combined With Fluoxetine in the Treatment of Depression
Brief Title: A Multicenter Clinical Study on Shuganjieyu Capsule Combined With Fluoxetine in the Treatment of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: Sichuan Jishengtang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Si Tianmei, Vice President of Institute of Mental Health, Peking University Sixth Hospital, Director of Research Laboratory on Psychopharmacology of Institute of Mental Health, Peking University Sixth Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V2.0
Record Dates: First submitted 2022-04-20; First posted 2022-05-04 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Outpatients / Inpatients With Depression
Keywords: Shuganjieyu capsule; depression
MeSH Terms: conditions — Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group: Shuganjieyu capsule (Experimental): Shuganjieyu capsule combined with Fluoxetine
  Interventions: Drug: Shuganjieyu capsule; Drug: Fluoxetine
- The control group: Shuganjieyu capsule simulator (Placebo Comparator): Fluoxetine monotherapy
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Shuganjieyu capsule — 2 capsules each time, twice per day. According to the study progress, the intervention can be adjusted to 4 capsules each time, twice per day
  Arms: The experimental group: Shuganjieyu capsule
Drug: Fluoxetine — Medication in basic study period: Fluoxetine (20 mg, once a day) Medication in the expanded study period: After 8 weeks of basic study period, if the reduction rate of HAMD-17 total scores is below 50 %, for the treatment group, the dosage of Fluoxetine will be adjusted to 40 mg / time, once a day.

SUMMARY:
This study mainly evaluates the efficacy and safety of Shuganjieyu capsule combined with Fluoxetine as well as the Fluoxetine monotherapy for the treatment of depression in the basic study, and also explores the efficacy for the extended study period as well as the efficacy and safety for the full trial period (basic study period and extended study period).

DETAILED DESCRIPTION:
Whole-course treatment serves as the principle for the treatment of depression, including symptom control in the acute phase, relapse prevention in the consolidation period and recurrence prevention in the maintenance period. Western medicine usually adopts antidepressant drugs combined with psychotherapy, mainly antidepressant SSRI at the current stage. It can selectively inhibit serotonin reuptake, so as to play an antidepressant role, but for somatic symptoms, the effect is general. Based on the overall regulation of body and mind, traditional Chinese medicine aims to achieve individualized treatment combing syndrome differentiation and treatment in a multi-channel, multi-target, and multi-level manner. At present, the combined application of antidepressant chemical drugs and Chinese patent medicines is complementary to each other from the perspective of mechanism and clinical practice. However, the study of Shuganjieyu capsule combined with antidepressant chemical drugs is mostly concentrated in the short term, and the benefits of long-term combined use of Shuganjieyu capsule remain to be further studied.

The purpose of this multicenter clinical study is to evaluate the efficacy and safety of Shuganjieyu capsule combined with Fluoxetine as well as the Fluoxetine monotherapy in the basic study period. Besides, the study aims to continue to observe the efficacy and safety in the extended study research period, so as to provide important clinical data for the whole-course medication.

Recruitment of outpatients / inpatients with depression. After screening the patients who met the inclusion criteria, the study collected demographic data, recorded symptoms and scale scores and improved relevant laboratory tests. The experimental group was treated with Shuganjieyu capsule combined with Fluoxetine, and the control group was treated with Fluoxetine. The related indexes were evaluated 2 ,4, 8, 12, 16 and 24 weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. In line with the diagnostic criteria for depression of Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5);
2. Age: 18-65 (including 18 and 65), gender unlimited;
3. Hamilton Rating Scale for Depression (HAMD-17) score≥18 in the screening period, and the 13th score≥2;
4. For women of childbearing age, pregnancy test must be negative and not in lactation. The contraception measure must be accepted by the Investigators. Participants should agree to maintain this measure throughout the whole process;
5. Sign the informed consent form voluntarily and agree to participate in all visits, examinations and treatment as required by the trial protocol.

Exclusion Criteria:

1. Treatment-resistant depression (patients with poor clinical efficacy of antidepressants with two or more different mechanisms after sufficient and full course of treatment);
2. Patients who meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia pedigree and other mental disorders, bipolar and related disorders, anxiety disorders, obsessive-compulsive and related disorders, somatic symptoms and related disorders);
3. Depression caused by psychoactive drugs;
4. Patients with severe suicide (HAMD-17 suicide score≥3) and injury tendency;
5. Patients with serious or unstable cardiovascular, cerebrovascular, liver, kidney, endocrine, digestive and blood diseases;
6. Depressive episodes secondary to other mental diseases or somatic diseases at an active stage;
7. ALT and AST values in the liver function examination are more than double the upper limit of reference value, or Scr value is above the upper limit of reference value;
8. Patients with a history of endocrine diseases such as hyperthyroidism and hypothyroidism who are currently active;
9. Patients who had undergone psychiatric surgery or electroconvulsive therapy in the past three months;
10. Anyone with an allergic constitution known or suspected to have an allergic history to Hypericum perforatum L., Eleutherococcus senticosus and Fluoxetine;
11. Those who have previously failed Shuganjieyu capsule or Fluoxetine treatment;
12. Women in pregnancy or lactation period. Women who plan to get pregnant during the study and within six months;
13. Patients with psychoactive substance abuse or dependence in the past 12 months;
14. Long-term use of caffeine and nicotine;
15. Patients who have received or are receiving any other clinical trial drug treatment within three months before the trial;
16. Patients who are taking drugs that interfere with the efficacy evaluation of the investigational drugs, and drugs that are forbidden to be used in combination with the test drugs. Patients who have received antidepressant drugs for systematical treatment within 4 weeks;
17. Those who are regarded as unsuitable by investigators for this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton depression rating scale (HAMD-17) total scores change | Day 0 to Day 56
  The change value of HAMD-17 total scores compared to the baseline (V1) after 8 weeks of treatment

SECONDARY OUTCOMES:
17-item Hamilton depression rating scale (HAMD-17) total scores change at early time points | Day 0 to Day 14, Day 0 to Day 28
  The change value of HAMD-17 total scores compared to the baseline
Hamilton anxiety rating scale (HAMA) total score change | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The change value of HAMA total scores compared to the baseline
Patient Health Questionnaire-15 (PHQ-15) score change | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The change value of PHQ-15 total scores compared to the baseline
Clinical Global Impression (CGI) score change | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The change value of CGI total scores compared to the baseline
Pittsburgh Sleep Quality Index (PSQI) score change | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The change value of PSQI total scores compared to the baseline
Dimensional Anhedonia Rating Scale (DARS) total score change | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The change value of DARS total scores compared to the baseline
Temporal Experience of Pleasure Scale (TEPS) total score change | Day 0 to Day 14, Day 0 to Day 28, Day 0 to Day 56
  The change value of TEPS total scores compared to the baseline
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) total score change | Day 0 to Day 56
  The change value of Q-LES-Q-SF total scores compared to the baseline

OTHER OUTCOMES:
17-item Hamilton depression rating scale (HAMD-17) change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change value of total score comared to the Week 8 time point
Relapse rate | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  When V4 shows clinical benefit after 8 weeks of treatment, the relapse rate of depression symptoms among participants after 12, 16, 24 weeks of treatment compared to V4 of 8-week treatment;
the rate of changing medicines | Day 56 to Day 168
  The rate of changing medicines among participants with 8 weeks of treatment when V4 entering the extended study period
Hamilton anxiety rating scale (HAMA) change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change value of total score comared to the Week 8 time point
Clinical Global Impression (CGI) score change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change comared to the Week 8 time point
Patient Health Questionnaire-15 (PHQ-15) score change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change comared to the Week 8 time point
Pittsburgh Sleep Quality Index (PSQI) score change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change comared to the Week 8 time point
Dimensional Anhedonia Rating Scale (DARS) total score change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change comared to the Week 8 time point
Temporal Experience of Pleasure Scale (TEPS) total score change in the extended period | Day 56 to Day 84, Day 56 to Day 112, Day 56 to Day 168
  The change comared to the Week 8 time point

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu
  - First Hospital, Shanxi Medical University, Taiyuan, Shanxi
  - Institute of Mental Health, Peking University Sixth Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No